CLINICAL TRIAL: NCT03228589
Title: The Effect of 8 Weeks Intake of a Probiotic Strain on a 6 Week Aspirin-induced Intestinal Deterioration Challenge in Healthy Volunteers - a Randomized, Double-blind, Placebo-controlled, Two Armed, Parallel Group Trial.
Brief Title: The Effect of a Probiotic Strain on Aspirin-induced GI Damage.
Acronym: PIP-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-GI-025
Record Dates: First submitted 2017-07-04; First posted 2017-07-25 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Side Effects of Acetylsalicylic Acid Use

STUDY DESIGN:
Intervention Model Description: Aspirin challenge model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic strain (Experimental): Active arm treated with the probiotic strain for 8 weeks.
  Interventions: Dietary Supplement: probiotic strain
- Placebo (Placebo Comparator): Placebo arm treated with placebo capsules (identical to active product capsule besides the bacteria) for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: probiotic strain — 8 weeks of treatment with probiotic strain
  Arms: probiotic strain
Dietary Supplement: Placebo — 8 weeks of treatment
  Arms: Placebo

SUMMARY:
This trial is a single-site, randomised, double-blind, placebo-controlled, two-armed, parallel-group trial in healthy, adult volunteers. The trial will investigate the effect of daily intake of a probiotic strain versus placebo when co-administered to daily intake of 300mg of Aspirin. The objective is to investigate the ability of the probiotic strain to attenuate and/or reverse Aspirin-induced deterioration of the small intestine.

DETAILED DESCRIPTION:
The trial includes a run-in period of two weeks duration followed by a six weeks intervention period where a probiotic strain/placebo and Aspirin is co-administered. After the 6 weeks, probiotic strain/placebo is given for two additional weeks to investigate the potential effects of the probiotic strain on intestinal healing after long-time Aspirin use.

Subjects will participate in the trial for a total duration of 10 weeks including the run-in phase. Besides the screening visit, the trial will consist of 6 visits.

After having given their written informed consent, subjects will complete screening procedures to evaluate their eligibility for participation in the trial and complete a run-in period of two weeks duration to washout possible pre-trial probiotics and/or use of medication. After baseline assessments at Visit 2, subjects will start daily intake of 300mg Aspirin and also be randomly assigned to 8 weeks daily intake of active or placebo product in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy and without any gastrointestinal discomfort/pain symptoms
* Age ≥ 18 - ≤ 40 years of both gender (aim of 1/3 of each gender in each arm)
* Sedentary lifestyle (weekly training load below 2 hours within endurance sports)
* Willing to abstain from any other probiotic products and/or medication known to alter gastrointestinal function throughout the participation of the trial

Exclusion Criteria:

* Abdominal surgery which, as judged by the investigator, might affect the GI function (except appendectomy and cholecystectomy)
* History of peptic ulcer disease
* Any known bleeding disorder
* Allergy to Aspirin
* History of H. pylori disease
* Resting diastolic blood pressure ≥ 90 mmHg
* Resting systolic blood pressure ≥ 140 mmHg
* A current diagnosis of psychiatric disease
* Systemic use of antibiotics, steroids (except contraceptives) or antimicrobial medication in the last 2 months
* BMI > 27
* Daily usage of non-steroidal anti-inflammatory drugs in the last 2 months or incidental use in the last 2 weeks prior to screening (Aspirin, Ibuprofen, Diclofenac, Naproxen, Celecoxib, Mefenamic acid, Etoricoxib, Indometacin)
* Usage of medications, except contraceptives, in the last 2 weeks prior to screening
* Diagnosed inflammatory gastrointestinal disease and/or irritable bowel syndrome
* Lactose intolerance
* Any other disease that, by the Investigators discretion, could interfere with the intestinal barrier function of the subject
* Participation in other clinical trials in the past 2 months prior to screening
* Regular use of probiotics in the last 2 months
* Smoking and/or frequent use of other nicotine products
* Desire and/or plans on changing current diet and/or exercise regime during the participation of this trial
* Use of laxatives, anti-diarrheals, anti-cholinergics and PPI within last 2 months prior to screening
* Use of immunosuppressant drugs within last 4 weeks prior to screening
* For Women: Pregnancy or lactation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Lewis score from capsule endoscopy | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on small intestinal mucosa damage when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve of the capsule endoscopy Lewis score between Visit 2 (randomization) and Visit 7 (end of treatment).

SECONDARY OUTCOMES:
Mucosal ulcer number | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on small intestinal mucosa damage when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve of the capsule endoscopy mucosal total ulcer number between Visit 2 (randomization) and Visit 7 (end of treatment).
Pain module score of the GSRS questionnaire | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on gastrointestinal symptoms when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve of pain module score of the GSRS questionnaire between Visit 2 (randomization) and Visit 7 (end of treatment).
Blood I-FABP concentration | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on small intestinal mucosa damage when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve for Visit 2-Visit 7 blood I-FABP concentration.
Total score of the GSRS questionnaire | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on gastrointestinal symptoms when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve of total score of the GSRS questionnaire between Visit 2 (randomization) and Visit 7 (end of treatment).
Mucosal red spots number | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on small intestinal mucosa damage when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve of the capsule endoscopy mucosal red spot number between Visit 2 (randomization) and Visit 7 (end of treatment).
Feces Calprotectin concentration. | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on small intestinal mucosa damage when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve for Visit 2-Visit 7 feces Calprotectin concentration.
blood Calprotectin concentration | 8 weeks
  The effect of 8 weeks oral supplementation of probiotic strain versus placebo on small intestinal mucosa damage when co-administered to a 6 week Aspirin challenge measured as the area-under-the-curve of the blood Calprotectin concentration between Visit 2 (randomization) and Visit 7 (end of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Buckley, Dr, Principal Investigator — GI Physiology Laboratory, Mercy University Hospital
Locations (1):
- Atlantia Food Clnical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortensen B, Murphy C, O'Grady J, Lucey M, Elsafi G, Barry L, Westphal V, Wellejus A, Lukjancenko O, Eklund AC, Nielsen HB, Baker A, Damholt A, van Hylckama Vlieg JET, Shanahan F, Buckley M. Bifidobacteriumbreve Bif195 Protects Against Small-Intestinal Damage Caused by Acetylsalicylic Acid in Healthy Volunteers. Gastroenterology. 2019 Sep;157(3):637-646.e4. doi: 10.1053/j.gastro.2019.05.008. Epub 2019 May 13. PMID 31095949